CLINICAL TRIAL: NCT00272727
Title: Improved Quality of the Treatment and Increased Compliance in Asthmatics Through the Dialog Tool Soren - Between Patient and Caregiver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NIS-RDK-DUM-2005/1; AZ-SOREN
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma; dialog tool; compliance
MeSH Terms: conditions — Asthma; Patient Compliance | interventions — Caregivers

INTERVENTIONS:
Behavioral: Dialog tool for caregivers

SUMMARY:
The purpose of the study is to assess if a dialog tool can improve compliance and asthma control in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma >/= 3 months,
* Prescribed daily use of inhaled glucocorticosteroid

Exclusion Criteria:

* Asthma exacerbation within the last month

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2006-02; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
ACQ

SECONDARY OUTCOMES:
Ability to follow prescription, AQLQ, lung function, No, eosinophil

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Denmark Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Copenhagen, Denmark